CLINICAL TRIAL: NCT06889896
Title: Clinical Evaluation of Blood-Based Assays for Rapid Detection of Aβ Pathology in Alzheimer's Disease
Acronym: CLEAR AD
Status: Enrolling by invitation | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024KY305
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer's Disease Diagnosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood plasma and blood cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- AD: There are clear complaints of cognitive impairment, and the diagnoses of AD meet the NIA-AA 2011 diagnostic criteria.
  Interventions: Diagnostic Test: After Blood samples collection, these samples are analyzed at a central laboratory under blinded conditions using multiple detection methods to measure plasma levels of Aβ40, Aβ42, t-tau, and p-tau
- MCI（Aβ PET+）: There are clear complaints of cognitive impairment, and the diagnoses of MCI meet the NIA-AA 2011 diagnostic criteria. Amyloid protein PET indicated positive within the last 3 months."
  Interventions: Diagnostic Test: After Blood samples collection, these samples are analyzed at a central laboratory under blinded conditions using multiple detection methods to measure plasma levels of Aβ40, Aβ42, t-tau, and p-tau
- MCI（Aβ PET-）: There are clear complaints of cognitive impairment, and the diagnoses of MCI meet the NIA-AA 2011 diagnostic criteria.Amyloid protein PET indicated negative within the last 3 months
  Interventions: Diagnostic Test: After Blood samples collection, these samples are analyzed at a central laboratory under blinded conditions using multiple detection methods to measure plasma levels of Aβ40, Aβ42, t-tau, and p-tau
- Non-AD dementia: Non-AD dementia is defined as patients who have a decline in cognitive abilities but are diagnosed with dementia due to other reasons (including but not limited to FTD, DLB, VD, PDD, etc.
  Interventions: Diagnostic Test: After Blood samples collection, these samples are analyzed at a central laboratory under blinded conditions using multiple detection methods to measure plasma levels of Aβ40, Aβ42, t-tau, and p-tau
- Cognitively normal controls: No complaints of cognitive impairment, scores within the normal range, and amyloid protein PET negative
  Interventions: Diagnostic Test: After Blood samples collection, these samples are analyzed at a central laboratory under blinded conditions using multiple detection methods to measure plasma levels of Aβ40, Aβ42, t-tau, and p-tau

INTERVENTIONS:
Diagnostic Test: After Blood samples collection, these samples are analyzed at a central laboratory under blinded conditions using multiple detection methods to measure plasma levels of Aβ40, Aβ42, t-tau, and p-tau — The CLEAR-AD study is an ongoing population-based cross-sectional study, currently recruiting 400 participants in ten centers in China. The study includes cognitively normal controls, individuals with mild cognitive impairment (MCI) - categorized as amyloid-positive and amyloid-negative - as well as patients with dementia, also divided into amyloid-positive and amyloid-negative groups. All participants undergo amyloid PET scans using tracers such as AV1, AV45, and PIB. Blood samples are collected within three months prior to the PET scan or from existing samples collected after January 1, 2024, that meet quality standards. After collection, these samples are analyzed at a central laboratory under blinded conditions using multiple detection methods to measure plasma levels of Aβ40, Aβ42, t-tau, and p-tau181/217. The detection technologies included single-molecule immunoassay, digital immunoassay chips, magnetic particle chemiluminescence, and flow cytometry fluorescence. The objective i

SUMMARY:
Background: Blood-based biomarkers show promise in predicting Alzheimer's disease (AD) pathology and progression; however, inconsistencies in detection standards hinder clinical application. A head-to-head comparison of commercially available biomarkers is crucial for optimizing the clinical pathway for AD screening and diagnosis.

Method: The CLEAR-AD study is an ongoing population-based cross-sectional study, currently recruiting 400 participants in ten centers in China. The study includes cognitively normal controls, individuals with mild cognitive impairment (MCI) - categorized as amyloid-positive and amyloid-negative - as well as patients with dementia, also divided into amyloid-positive and amyloid-negative groups. All participants undergo amyloid PET scans using tracers such as AV1, AV45, and PIB. Blood samples are collected within three months prior to the PET scan or from existing samples collected after January 1, 2024, that meet quality standards. After collection, these samples are analyzed at a central laboratory under blinded conditions using multiple detection methods to measure plasma levels of Aβ40, Aβ42, t-tau, and p-tau181/217. The detection technologies included single-molecule immunoassay, digital immunoassay chips, magnetic particle chemiluminescence, and flow cytometry fluorescence. The objective is to assess the sensitivity and specificity of different plasma biomarker levels in predicting amyloid pathology confirmed by Aβ-PET.

Result: The study uses Aβ-PET as the reference standard to evaluate the sensitivity and specificity of various AD plasma biomarkers across different detection methods in diagnosing amyloid pathology. The analysis included generating receiver operating characteristic (ROC) curves, determining optimal cut-off values, and developing a predictive model that integrates multiple biomarker parameters and clinical data. Results is considered statistically significant with a p-value of less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

Patient Group (including MCI, AD, and Non-AD Dementia):

1. Clear complaints of cognitive impairment, with MCI and AD diagnoses meeting the NIA-AA 2011 diagnostic criteria. Non-AD dementia is defined as patients with cognitive decline diagnosed with dementia due to other reasons (including but not limited to FTD, DLB, VD, PDD, etc.).
2. Able to provide informed consent or have a legal guardian who can sign the consent form.
3. Completed a full set of cognitive assessments, including MMSE and CDR.
4. Able to provide a history of chronic diseases, including cardiovascular diseases, diabetes, etc., and medication history.
5. Have undergone amyloid protein PET scans that meet the quality requirements of this study (tracers PiB, AV1, or AV45), and can provide original imaging data for quantitative analysis without conflict.
6. Can provide frozen plasma from a biobank collected after January 1, 2024, with a time interval of ≤3 months from the amyloid protein PET scan. If no frozen plasma is available, willing to provide an additional 5ml of whole blood for biomarker testing in this project. The process of blood collection, plasma separation, storage, and transportation meets the quality requirements of this study (see blood testing SOP).
7. Have 3D-T1 structural MRI images taken within 3 months before and after the amyloid protein PET scan and can provide original imaging data without conflict.

Normal Control Group:

1. Subjects with a CDR score of 0 and who have undergone amyloid protein PET scans that are negative.
2. Able to provide informed consent.
3. Completed a full set of cognitive assessments, including MMSE and CDR.
4. Able to provide a history of chronic diseases, including cardiovascular diseases, diabetes, etc., and medication history.
5. Have undergone amyloid protein PET scans that meet the quality requirements of this study (tracers PiB, AV1, or AV45), and can provide original imaging data for quantitative analysis without conflict.
6. Can provide frozen plasma from a biobank collected after January 1, 2024, with a time interval of ≤3 months from the amyloid protein PET scan. If no frozen plasma is available, willing to provide an additional 5ml of whole blood for biomarker testing in this project. The process of blood collection, plasma separation, storage, and transportation meets the quality requirements of this study (see blood testing SOP).
7. Have 3D-T1 structural MRI images taken within 3 months before and after the amyloid protein PET scan and can provide original imaging data without conflict.

Exclusion Criteria:

1. History of Mental Illness:** Depression (Geriatric Depression Scale [GDS] > 7 points or Hamilton Depression Rating Scale [17-item version] > 7 points);
2. History of Central Nervous System Diseases:** Including infections, epilepsy, multiple sclerosis, toxic metabolic diseases, familial hereditary diseases, neurotumors, etc.;
3. Severe Stroke Sequelae:** mRS > 3 points or a documented history of stroke sequelae;
4. Severe Liver and Kidney Dysfunction at Diagnosis:** ALT ≥ 5 times the upper limit of normal, or estimated glomerular filtration rate (eGFR) < 30 ml·min-¹·(1.73 m²)-¹, or patients requiring renal replacement therapy;
5. History of Drug Abuse and Severe Alcoholism;**
6. Prior Use of Anti-Aβ or Other Disease-Modifying Treatments,** unless there is clear evidence of a placebo group;
7. Severe Hyperlipidemia:** Triglycerides ≥ 5.6 mmol/L or visible chylomicron changes in plasma.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The CLEAR-AD study is an ongoing population-based cross-sectional study, currently recruiting 400 participants in ten centers in China. The study includes cognitively normal controls, individuals with mild cognitive impairment (MCI) - categorized as amyloid-positive and amyloid-negative - as well as patients with dementia, also divided into amyloid-positive and amyloid-negative groups. All participants undergo amyloid PET scans using tracers such as AV1, AV45, and PIB.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the sensitivity and specificity of blood biomarkers in predicting amyloid pathology confirmed by Aβ-PET under different testing methods | 2025.08

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, The First Affiliated Hospital of USTC, Division of Life Sciences and Medicine, University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
All interested researchers can obtain relevant information through the contact details of the researchers